CLINICAL TRIAL: NCT05718544
Title: Effect of Mini-dose Esketamine-dexmedetomidine Supplemented Analgesia on Long-term Outcomes Following Scoliosis Correction Surgery: 2-year Follow-up of a Randomized Controlled Trial
Brief Title: Mini-dose Esketamine-dexmedetomidine Supplemented Analgesia and Long-term Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-017
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Scoliosis Correction; Postoperative Analgesia; Esketamine; Dexmedetomidine; Chronic Postsurgical Pain
Keywords: Scoliosis Correction; Postoperative analgesia; Esketamine; Dexmedetomidine; Chronic Postsurgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Esketamine; Dexmedetomidine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined supplement (Experimental): Patient-controlled analgesia is established with esketamine 50 mg, dexmedetomidine 200 microgram, and sufentanil 4 microgram/kg (maximum 250 microgram), diluted with normal saline to 200 ml, and programmed to administer 2-ml boluses with a lockout interval of 8 minutes and a background infusion rate at 1 ml/h.
  Interventions: Drug: Esketamine; Drug: Dexmedetomidine; Drug: Sufentanil
- Placebo (Placebo Comparator): Patient-controlled analgesia is established with sufentanil 4 microgram/kg (maximum 250 microgram), diluted with normal saline to 200 ml, and programmed to administer 2-ml boluses with a lock-out interval of 8 minutes and a background infusion rate at 1 ml/h.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Esketamine — Esketamine 50 mg is included in the mixture for patient-controlled analgesia.
  Arms: Combined supplement
Drug: Dexmedetomidine — Dexmedetomidine 200 microgram is included in the mixture for patient-controlled analgesia.
  Arms: Combined supplement
Drug: Sufentanil — Sufentanil 4 microgram/kg (maximum 250 microgram) is included in the mixture for patient-controlled analgesia.

SUMMARY:
Chronic postsurgical pain (CPSP) refers to pain that occurs or increases after surgery and lasts longer than 3 months. Severe postoperative acute pain is one of the major risk factors of CPSP. Spine surgery brings severe postoperative pain due to large trauma and long duration. Ketamine and esketamine are N-methyl-D-aspartate receptor antagonists; they have anti-hyperalgesic effects and may reduce CPSP. Dexmedetomidine is an alpha 2-adrenoceptor agonist with sedative, anxiolytic, and analgesic effect; it is frequently used as an adjuvant to postoperative analgesia. In a previous trial of the investigators, 200 patients following scoliosis correction surgery were randomzied to receive opioid analgsia supplemented with either mini-dose esketamine-dexmedetomidine combination or placebo. The results showed that esketamine-dexmedetomidine supplement analgesia significantly improved analgesia and sleep quality after surgery. This study is designed to test the hypothesis that mini-dose esketamine-dexmedetomidine supplemented analgesia may reduce CPSP at 2 years after scoliosis correction surgery.

DETAILED DESCRIPTION:
Chronic postsurgical pain (CPSP) refers to pain that occurs or increases after surgery and lasts longer than 3 months. Pain can be limited to the surgical area or projected to the innervated area. The incidence of CPSP is about 10-50%, and the incidence of moderate to severe CPSP is as high as 11.8%. The risk factors of CPSP include severe postoperative acute pain, long duration surgery, and related nerve injury. Spine surgery brings severe lesion and postoperative pain due to large trauma and long duration, with a median pain score of 7 (interquaritle range, 4 to 8) on the first day after surgery. And the incidence of persistent pain is as high as 75%.

Ketamine is a non-competitive N-methyl-D-aspartate (NMDA) receptor antagonists. NMDA receptors are located in the brain and spinal cord of the central nervous system, responsible for the afferent of noxious stimuli. After nerve injury, the continuous activity and transmission of nociceptive signals up-regulates NMDA receptors in the dorsal horn of the spinal cord, amplify the pain signal to the brain, which may be related to the pathogenesis of CPSP. Ketamine has anti-hyperalgesia effects and may reduce the occurrence of CPSP by blocking NMDA receptors. Esketamine is the S-enantiomer of racemic ketamine with stronger analgesic effect and lower incidence of adverse reactions. In previous studies, opioid-dependent patients who received low-dose ketamine/esketamine infusion during the perioperative period had decreased pain scores and opioid requirement at 6 weeks, 6 months, and 1 year after surgery. However, results of patients without opioid dependence are controversial. In addition, ketamine/esketamine are approved for refractory depression. There is a significant correlation between anxiety/depression and chronic pain. This may also be one of the mechanisms in preventing CPSP.

Dexmedetomidine is a highly selective α2 receptor agonist with sedative, anxiolytic, and analgesic effects. It can improve analgesic effect, reduce opioid consumption, and reduce opioid-related adverse reactions when used in the perioperative period. Meanwhile, dexmedetomidine can prolong total sleep time, improve sleep efficiency, and increase subjective sleep quality, possibly by activating the endogenous sleep pathway. The sedative effect of dexmedetomidine may help to reduce the psychiatric adverse reactions of ketamine. However, data is lacking regarding the effect of dexmedetomidine on chronic postsurgical pain.

In a previous trial of the investigators, 200 patients following scoliosis correction surgery were randomzied to receive opioid analgsia supplemented with either mini-dose esketamine-dexmedetomidine combination or placebo. The results showed that esketamine-dexmedetomidine supplement analgesia significantly reduced the incidence of moderate and severe pain and improved the quality of sleep during the perioperative period; adverse reactions were not significantly increased (unpublished data). This study is designed to test the hypothesis that mini-dose esketamine-dexmedetomidine supplemented analgesia may reduce CPSP at 2 years after scoliosis correction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years;
* Scheduled for scoliosis correction surgery;
* Required patient-controlled intravenous analgesia (PCIA) after surgery.

Exclusion Criteria:

* Preoperative sick sinus syndrome, severe sinus bradycardia (heart rate <50 beats per minute), atrioventricular block grade II or above without pacemaker, congenital heart disease, arrhythmia, or other serious cardiovascular diseases with a New York Heart Association class ≥III;
* Obstructive sleep apnea syndrome, or a STOP-Bang score ≥3 in combination with a serum bicarbonate level ≥28 mmol/L;
* Comorbid hyperthyroidism or pheochromocytoma;
* History of schizophrenia, epilepsy, myasthenia gravis;
* Preoperative delirium or communication barrier;
* Severe liver dysfunction (Child-Pugh grade C), severe renal dysfunction (preoperative dialysis), or American Society of Anaesthesiologists grade ≥IV;
* Body weight <40 kg;
* Enrolled in other clinical studies;
* Loss to follow-up;
* Other conditions that were considered unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Incidence of chronic postsurgical pain at 2 years after surgery | At 2 years after surgery
  Chronic postsurgical pain (CPSP) is defined as pain persisted for at least three months after surgery, that is not present before surgery or that has different characteristics, and other possible causes of the pain are excluded (e.g., cancer recurrence, infection).

SECONDARY OUTCOMES:
Severity of chronic pain at 2 years after surgery | At 2 years after surgery
  Severity of chronic pain is assessed with the Brief Pain Inventory (BPI). The BPI gives two main scores: a pain severity score and a pain interference score. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40.
Interference of chronic pain at 2 years after surgery | At 2 years after surgery
  Interference of chronic pain is assessed with the Brief Pain Inventory (BPI). The BPI gives two main scores: a pain severity score and a pain interference score. The pain interference score corresponds to the item on pain interference. The seven subitems are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70.
Proportion of chronic analgesic use after surgery | Up to 2 years after surgery
  Chronic analgesic use is defined as consecutive use of analgesics for more than 3 months.
Proportion of analgesic use at 2 years after surgery | At 2 years after surgery
  Proportion of analgesic use at 2 years after surgery (consecutive use of analgesics for more than 1 week within 3 months).
Subjective sleep quality at 2 years after surgery | At 2 years after surgery
  Subjective sleep quality at 2 years is assessed with the Pittsburgh Sleep Quality Index (PSQI). PSQI is a 7-item questionnaire consisting 19 self-rated questions that assesses sleep quality over the last month, each weighted equally on a 0-3 scale; higher scores indicate worse sleep quality.
Depression severity at 2 years after surgery | At 2 years after surgery
  Depression is assessed with the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 includes 9-item requiring responses of 0 (not at all) to 3 (nearly every day) to assess the occurrence of depressive symptoms over the last two weeks. It has 8 items on depressive symptoms and 1 focused on suicidal ideation. Total scores range from 0 to 27, with higher score indicating more severe symptoms.
Quality of life at 2 years after surgery | At 2 years after surgery
  Quality of life is assessed using the Scoliosis Research Society-22 (SRS-22) patient questionnaire, which consists of five domains: function, pain, mental health, self-image, and satisfaction with management.
Event-free survival | Up to 2 years after surgery
  Event indicates any condition that requires hospitalization and clinical treatment for unexpected reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willis DE, Goldstein PA. Targeting Affective Mood Disorders With Ketamine to Prevent Chronic Postsurgical Pain. Front Pain Res (Lausanne). 2022 Jun 27;3:872696. doi: 10.3389/fpain.2022.872696. eCollection 2022. PMID 35832728
- [Background] Fletcher D, Stamer UM, Pogatzki-Zahn E, Zaslansky R, Tanase NV, Perruchoud C, Kranke P, Komann M, Lehman T, Meissner W; euCPSP group for the Clinical Trial Network group of the European Society of Anaesthesiology. Chronic postsurgical pain in Europe: An observational study. Eur J Anaesthesiol. 2015 Oct;32(10):725-34. doi: 10.1097/EJA.0000000000000319. PMID 26241763
- [Background] Wylde V, Dennis J, Beswick AD, Bruce J, Eccleston C, Howells N, Peters TJ, Gooberman-Hill R. Systematic review of management of chronic pain after surgery. Br J Surg. 2017 Sep;104(10):1293-1306. doi: 10.1002/bjs.10601. Epub 2017 Jul 6. PMID 28681962
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Hussain A, Erdek M. Interventional pain management for failed back surgery syndrome. Pain Pract. 2014 Jan;14(1):64-78. doi: 10.1111/papr.12035. Epub 2013 Feb 3. PMID 23374545
- [Background] Dunn LK, Yerra S, Fang S, Hanak MF, Leibowitz MK, Tsang S, Durieux ME, Nemergut EC, Naik BI. Incidence and Risk Factors for Chronic Postoperative Opioid Use After Major Spine Surgery: A Cross-Sectional Study With Longitudinal Outcome. Anesth Analg. 2018 Jul;127(1):247-254. doi: 10.1213/ANE.0000000000003338. PMID 29570151
- [Background] Leider HL, Dhaliwal J, Davis EJ, Kulakodlu M, Buikema AR. Healthcare costs and nonadherence among chronic opioid users. Am J Manag Care. 2011 Jan;17(1):32-40. PMID 21348566
- [Background] Agarwal D, Chahar P, Chmiela M, Sagir A, Kim A, Malik F, Farag E. Multimodal Analgesia for Perioperative Management of Patients presenting for Spinal Surgery. Curr Pharm Des. 2019;25(19):2123-2132. doi: 10.2174/1381612825666190708174639. PMID 31298146
- [Background] Bartova L, Papageorgiou K, Milenkovic I, Dold M, Weidenauer A, Willeit M, Winkler D, Kasper S. Rapid antidepressant effect of S-ketamine in schizophrenia. Eur Neuropsychopharmacol. 2018 Aug;28(8):980-982. doi: 10.1016/j.euroneuro.2018.05.007. Epub 2018 Jul 2. PMID 30041987
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Am J Psychiatry. 2018 Jul 1;175(7):620-630. doi: 10.1176/appi.ajp.2018.17060720. Epub 2018 Apr 16. PMID 29656663
- [Background] Segmiller F, Ruther T, Linhardt A, Padberg F, Berger M, Pogarell O, Moller HJ, Kohler C, Schule C. Repeated S-ketamine infusions in therapy resistant depression: a case series. J Clin Pharmacol. 2013 Sep;53(9):996-8. doi: 10.1002/jcph.122. Epub 2013 Jul 24. No abstract available. PMID 23893490
- [Background] Loftus RW, Yeager MP, Clark JA, Brown JR, Abdu WA, Sengupta DK, Beach ML. Intraoperative ketamine reduces perioperative opiate consumption in opiate-dependent patients with chronic back pain undergoing back surgery. Anesthesiology. 2010 Sep;113(3):639-46. doi: 10.1097/ALN.0b013e3181e90914. PMID 20693876
- [Background] Nielsen RV, Fomsgaard JS, Siegel H, Martusevicius R, Nikolajsen L, Dahl JB, Mathiesen O. Intraoperative ketamine reduces immediate postoperative opioid consumption after spinal fusion surgery in chronic pain patients with opioid dependency: a randomized, blinded trial. Pain. 2017 Mar;158(3):463-470. doi: 10.1097/j.pain.0000000000000782. PMID 28067693
- [Background] Nielsen RV, Fomsgaard JS, Nikolajsen L, Dahl JB, Mathiesen O. Intraoperative S-ketamine for the reduction of opioid consumption and pain one year after spine surgery: A randomized clinical trial of opioid-dependent patients. Eur J Pain. 2019 Mar;23(3):455-460. doi: 10.1002/ejp.1317. Epub 2018 Oct 14. PMID 30246357
- [Background] Nielsen RV. Adjuvant analgesics for spine surgery. Dan Med J. 2018 Mar;65(3):B5468. PMID 29510816
- [Background] Carley ME, Chaparro LE, Choiniere M, Kehlet H, Moore RA, Van Den Kerkhof E, Gilron I. Pharmacotherapy for the Prevention of Chronic Pain after Surgery in Adults: An Updated Systematic Review and Meta-analysis. Anesthesiology. 2021 Aug 1;135(2):304-325. doi: 10.1097/ALN.0000000000003837. PMID 34237128
- [Background] Giusti EM, Lacerenza M, Gabrielli S, Manzoni GM, Manna C, D'Amario F, Marcacci M, Castelnuovo G. Psychological factors and trajectories of post-surgical pain: A longitudinal prospective study. Pain Pract. 2022 Feb;22(2):159-170. doi: 10.1111/papr.13074. Epub 2021 Sep 25. PMID 34498384
- [Background] Peng K, Zhang J, Meng XW, Liu HY, Ji FH. Optimization of Postoperative Intravenous Patient-Controlled Analgesia with Opioid-Dexmedetomidine Combinations: An Updated Meta-Analysis with Trial Sequential Analysis of Randomized Controlled Trials. Pain Physician. 2017 Nov;20(7):569-596. PMID 29149140
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Hong H, Zhang DZ, Li M, Wang G, Zhu SN, Zhang Y, Wang DX, Sessler DI. Impact of dexmedetomidine supplemented analgesia on delirium in patients recovering from orthopedic surgery: A randomized controlled trial. BMC Anesthesiol. 2021 Sep 13;21(1):223. doi: 10.1186/s12871-021-01441-3. PMID 34517840
- [Background] Zhang ZF, Su X, Zhao Y, Zhong CL, Mo XQ, Zhang R, Wang K, Zhu SN, Shen YE, Zhang C, Wang DX. Effect of mini-dose dexmedetomidine supplemented intravenous analgesia on sleep structure in older patients after major noncardiac surgery: A randomized trial. Sleep Med. 2023 Feb;102:9-18. doi: 10.1016/j.sleep.2022.12.006. Epub 2022 Dec 20. PMID 36587547
- [Background] Hu ZC, Xu G, Zhang XW, Ma K, Jin JJ, Li PS. [Meta-analysis of the effects of dexmedetomidine combined with ketamine during dressing changes in burn patients]. Zhonghua Shao Shang Za Zhi. 2020 Jun 20;36(6):458-464. doi: 10.3760/cma.j.cn501120-20190327-00145. Chinese. PMID 32594705
- [Background] Lee KH, Lee SJ, Park JH, Kim SH, Lee H, Oh DS, Kim YH, Park YH, Kim H, Lee SE. Analgesia for spinal anesthesia positioning in elderly patients with proximal femoral fractures: Dexmedetomidine-ketamine versus dexmedetomidine-fentanyl. Medicine (Baltimore). 2020 May;99(20):e20001. doi: 10.1097/MD.0000000000020001. PMID 32443302
- [Background] Cheung KM, Senkoylu A, Alanay A, Genc Y, Lau S, Luk KD. Reliability and concurrent validity of the adapted Chinese version of Scoliosis Research Society-22 (SRS-22) questionnaire. Spine (Phila Pa 1976). 2007 May 1;32(10):1141-5. doi: 10.1097/01.brs.0000261562.48888.e3. PMID 17471100
- [Background] Li M, Wang CF, Gu SX, He SS, Zhu XD, Zhao YC, Zhang JT. Adapted simplified Chinese (mainland) version of Scoliosis Research Society-22 questionnaire. Spine (Phila Pa 1976). 2009 May 20;34(12):1321-4. doi: 10.1097/BRS.0b013e31819812b7. PMID 19455008